CLINICAL TRIAL: NCT00722826
Title: MRI Assessment of Right Ventricular Function in Patients After Repair of Tetralogy of Fallot
Brief Title: Tetralogy of Fallot Seed Grant
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H627-29142-02; UCSF Seed Grant FWA #00000068
Record Dates: First submitted 2008-07-23; First posted 2008-07-28 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Pulmonary Regurgitation After Repair of Tetralogy of Fallot
Keywords: Pulmonary Regurgitation; Tetralogy of Fallot
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with pulmonary regurgitation after surgical correction of ToF over 13 years old will be recruited from the UCSF adult congenital heart disease clinic. Since there is no data in the literature describing the prevalence of abnormal MRI volumetric and functional parameters in asymptomatic patients with PR after ToF repair, a pilot study with 30 patients will be conducted. Increase in sample size may be necessary in the future to accurately interpret the data. After informed consent is obtained, clinical history and physical examination as well as review of old charts will be performed to characterize these patient's clinical status. All patients will undertake a graduated supine bicycle exercise test with MVO2 measurement to assess exercise capacity.

MRI studies will be performed in a 1.5 tesla unit. SSFP cine images will be obtained in the short-axis plane encompassing the entire heart. Velocity-encoded cine MR images will be obtained perpendicular to the direction of blood flow in the main pulmonary artery. Volumetric and flow analysis will be performed in a separate dedicated workstation by a radiologist. End-diastolic volume, end-systolic volume, ejection fraction, total ejection fraction and pulmonary regurgitant fraction will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Patients over 13 years of age with pulmonary regurgitation after surgical correction of tetralogy of Fallot.

1. Adult patients with pulmonary regurgitation after surgical repair of tetralogy of Fallot who are under follow-up at the adult congenital heart disease clinic at UCSF or
2. Pediatric patients with pulmonary regurgitation after surgical repair of tetralogy of Fallot who are under follow-up at the pediatric congenital heart disease clinic at UCSF and are referred for a clinically indicated cardiac MRI studies or
3. Adult and pediatric patients with pulmonary regurgitation after surgical repair of tetralogy of Fallot who are referred for clinically indicated MRI studies at UCSF.

Exclusion Criteria:

Contraindication for MRI study. Claustrophobia.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a cross sectional study. Patients with pulmonary regurgitation after repair of tetralogy of Fallot assisted in the adult or pediatric congenital heart disease clinic or referred for clinical MRI studies at our institution will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Higgins, MD, Principal Investigator — UCSF Department of Radiology
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Geva T, Sandweiss BM, Gauvreau K, Lock JE, Powell AJ. Factors associated with impaired clinical status in long-term survivors of tetralogy of Fallot repair evaluated by magnetic resonance imaging. J Am Coll Cardiol. 2004 Mar 17;43(6):1068-74. doi: 10.1016/j.jacc.2003.10.045. PMID 15028368
- [Background] Davlouros PA, Kilner PJ, Hornung TS, Li W, Francis JM, Moon JC, Smith GC, Tat T, Pennell DJ, Gatzoulis MA. Right ventricular function in adults with repaired tetralogy of Fallot assessed with cardiovascular magnetic resonance imaging: detrimental role of right ventricular outflow aneurysms or akinesia and adverse right-to-left ventricular interaction. J Am Coll Cardiol. 2002 Dec 4;40(11):2044-52. doi: 10.1016/s0735-1097(02)02566-4. PMID 12475468
- [Background] Helbing WA, de Roos A. Clinical applications of cardiac magnetic resonance imaging after repair of tetralogy of Fallot. Pediatr Cardiol. 2000 Jan-Feb;21(1):70-9. doi: 10.1007/s002469910009. PMID 10672616
- [Background] Araoz PA, Reddy GP, Higgins CB. Congenital heart disease. In: Higgins CB, de Roos A, eds. Cardiovascular MRI and MRA. 1 ed. Philadelphia: Lippincott Williams & Wilkins, 2003; 122-135.
- [Background] Higgins CB, Caputo GR. Role of MR imaging in acquired and congenital cardiovascular disease. AJR Am J Roentgenol. 1993 Jul;161(1):13-22. doi: 10.2214/ajr.161.1.8517291.
- [Background] van der Geest RJ, Reiber JH. Quantification in cardiac MRI. J Magn Reson Imaging. 1999 Nov;10(5):602-8. doi: 10.1002/(sici)1522-2586(199911)10:53.0.co;2-c. PMID 10548768
- [Background] Higgins CB, Sakuma H. Heart disease: functional evaluation with MR imaging. Radiology. 1996 May;199(2):307-15. doi: 10.1148/radiology.199.2.8668769.
- [Background] Pettigrew RI, Oshinski JN, Chatzimavroudis G, Dixon WT. MRI techniques for cardiovascular imaging. J Magn Reson Imaging. 1999 Nov;10(5):590-601. doi: 10.1002/(sici)1522-2586(199911)10:53.0.co;2-s. PMID 10548767